CLINICAL TRIAL: NCT00116415
Title: Daily Antiretroviral Therapy (DART 1): An Open-Label, Single-Arm, Prospective, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Didanosine Enteric Coated (Ddl-EC) in Combination With Lamivudine (3TC) and Efavirenz (EFV) Once Daily in Anti-Retroviral Therapy (ART) Naive HIV-Infected Patients
Brief Title: DART I - A Phase IV Study of 3 Antiretroviral Medicines in Combination, in HIV Patients Who Have Not Been Previously Treated With Antiretroviral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI266-071
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections; AIDS
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — efavirenz; Didanosine; Lamivudine

INTERVENTIONS:
Drug: efavirenz; didanosine EC; lamivudine

SUMMARY:
The purpose of this study is to evaluate whether a therapy with an all once daily regimen of efavirenz (EFV), didanosine (ddI)-EC and lamivudine (3TC) leads to improved outcomes, as measured by viral load, CD4 counts, adherence, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older infected with HIV and weigh at least 40 kg.
* Plasma HIV RNA viral load of 1000 copies/mL or greater and CD4 count of 100 cells/mL or greater
* Be willing to use two forms of contraception throughout study
* No previous exposure to antiretroviral (ARV) drugs

Exclusion Criteria:

* Pregnancy or breastfeeding
* Physical or psychiatric disability
* Proven or suspected acute hepatitis within 30 days prior to study entry
* Active AIDS-defining opportunistic infection or disease
* History of acute or chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2002-03; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Estimate efficacy of ddI-EC/3TC/EFV given QD determined by proportion of patients with plasma HIV-1 RNA <400 copies/mL at 48 weeks

SECONDARY OUTCOMES:
Evaluate proportion of patients with plasma HIV RNA <400 copies/mL at Weeks 24, 48, 72, and 96.
Evaluate proportion of patients with plasma HIV RNA <50 copies/mL at Weeks 24, 48, 72, and 96
Determine viral suppression of plasma HIV RNA from change in baseline at week 48
Determine proportion of patients whose HIV viral load doesn't drop to undetectable level within 24 weeks
Evaluate time to undetectable plasma HIV RNA
Evaluate proportion of patients demonstrating virologic breakthrough
Evaluate proportion of patients demonstrating virologic failure
Evaluate time to virologic breakthrough and virologic failure
Measure magnitude and durability of changes in CD4 cell counts
Evaluate patient adherence with QD regimen using pill counts and AMAF
Determine pattern and emergence of HIV genotype resistance mutations in patients experiencing virologic failure
Explore QoL changes using MOS-HIV health survey
Evaluate safety and tolerability of QD regimen

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (9):
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Orlando, Florida
  - Local Institution, Columbus, Georgia
  - Local Institution, Boston, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Kansas City, Missouri
  - Local Institution, Hillsborough, New Jersey
  - Local Institution, The Bronx, New York
  - Local Institution, Dallas, Texas

REFERENCES:
- [Derived] Jayaweera D, Dejesus E, Nguyen KL, Grimm K, Butcher D, Seekins DW. Virologic suppression, treatment adherence, and improved quality of life on a once-daily efavirenz-based regimen in treatment-Naive HIV-1-infected patients over 96 weeks. HIV Clin Trials. 2009 Nov-Dec;10(6):375-84. doi: 10.1310/hct1006-375. PMID 20133268
- [Derived] Nunes EP, Santini de Oliveira M, Mercon M, Zajdenverg R, Faulhaber JC, Pilotto JH, Ribeiro JE, Norton M, Schechter M. Monotherapy with Lopinavir/Ritonavir as maintenance after HIV-1 viral suppression: results of a 96-week randomized, controlled, open-label, pilot trial (KalMo study). HIV Clin Trials. 2009 Nov-Dec;10(6):368-74. doi: 10.1310/hct1006-368. PMID 20133267